CLINICAL TRIAL: NCT03670758
Title: Protein S Activity in Women With Unexplained Infertility
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Esraa Gamal Ahmed (Other)
Collaborators: Ain Shams Maternity Hospital (Other)
Responsible Party: Sponsor-Investigator, Esraa Gamal Ahmed, Esraa Gamal Ahmed, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: AinShamsMH EAhmed
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Unexplained Female Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Will include 30 women with unexplained primary infertility; will be recruited from the outpatient infertility clinic
  Interventions: Diagnostic Test: Protein S activity
- Group 2: another 30 fertile women who got pregnant and delivered at least once in the previous year with no history of recurrent abortions; will recruited from outpatient gynecology clinic as control
  Interventions: Diagnostic Test: Protein S activity

INTERVENTIONS:
Diagnostic Test: Protein S activity — Intravenous blood sample

SUMMARY:
This study will add:

Finding out an association between Protein S activity and unexplained female infertility.

Aim:

Study hypothesis:

In women with unexplained infertility protein S activity may be low.

Study question:

In women with unexplained infertility does protein S activity low?.

This study aims to assess the activity of protein S activity in women with unexplained infertility.

Objectives:

The main objective of this study is:

To determine the prevalence of Protein S activity with unexplained female infertility and to compare its prevalence in fertile women among women attending outpatient clinics at Ain Shams University Maternity Hospital.

DETAILED DESCRIPTION:
1. Type of Study: Case Control Study.
2. Study Setting: Ain Shams University Maternity Hospital: outpatient Infertility clinic and outpatient gynecology clinic.
3. Study Population: The study will include women with unexplained infertility (Group 1; cases) and fertile women who got pregnant and delivered at least once in the previous year with no history of recurrent abortions nor history of secondary infertility (Group 2; control).

Group 1: Will include 30 women with unexplained primary infertility; will be recruited from the outpatient infertility clinic.

Group 2; another 30 fertile women who got pregnant and delivered at least once in the previous year with no history of recurrent abortions; will recruited from outpatient gynecology clinic as control.

According to inclusion and exclusion criteria listed below.

Inclusion criteria:

1. Age: 18 - 35 years old.
2. Normal husband's semen analysis, (WHO criteria):

   1. Count ≥ 15 million/ml.
   2. Motility: ≥ 40%
   3. Morphology: ≥ 4% normal morphology.
3. Documented ovulation.
4. Normal Follicle Stimulating Hormone, Luteinizing Hormone, Thyroid Stimulating Hormone, serum prolactin.
5. Patent Fallopian tubes.
6. Normal uterine cavity.

Exclusion criteria:

1. Patients aged less than 18 years or more than 35 years old.
2. Secondary infertility
3. Presence of male factor infertility
4. Anovulatory cycles.
5. Tubal block; Tubal disease is an important cause of infertility and should be speciﬁcally excluded.
6. Medical disorder that might affect pregnancy (e.g.: Diabetes, Thyroid dysfunction)
7. Patients with recurrent abortion.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 - 35 years old.
2. Normal husband's semen analysis, (WHO criteria):

   1. Count ≥ 15 million/ml.
   2. Motility: ≥ 40%
   3. Morphology: ≥ 4% normal morphology.
3. Documented ovulation.
4. Normal Follicle Stimulating Hormone, Luteinizing Hormone, Thyroid Stimulating Hormone, serum prolactin.
5. Patent Fallopian tubes.
6. Normal uterine cavity.

   -

Exclusion Criteria:

1. Patients aged less than 18 years or more than 35 years old.
2. Secondary infertility
3. Presence of male factor infertility
4. Anovulatory cycles.
5. Tubal block; Tubal disease is an important cause of infertility and should be speciﬁcally excluded.
6. Medical disorder that might affect pregnancy (e.g.: Diabetes, Thyroid dysfunction)
7. Patients with recurrent abortion. -

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study will include women with unexplained infertility
Study Population: The study will include women with unexplained infertility (Group 1; cases) and fertile women who got pregnant and delivered at least once in the previous year with no history of recurrent abortions nor history of secondary infertility (Group 2; control).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-09-05 (Estimated); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Estimated)

PRIMARY OUTCOMES:
Protein S activity | six months
  venous blood sample